CLINICAL TRIAL: NCT06005454
Title: The Impact of Fish Oil Supplementation on the Outcome of Children with Pneumonia in the Intensive Care Unit
Brief Title: The Impact of Fish Oil Supplementation on the Outcome of Children with Pneumonia I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Atef Abdelsattar Ibrahim, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-369-2022
Record Dates: First submitted 2023-08-10; First posted 2023-08-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Children with Pneumonia in intensive care unit receiving fish oil and the standard treatment (Experimental)
  Interventions: Dietary Supplement: Fish oil (Omega)
- Children with Pneumonia in intensive care unit receiving the standard treatment only (No Intervention)

INTERVENTIONS:
Dietary Supplement: Fish oil (Omega) — We will use a dietary supplement source of omega 3 fatty acids from the available syrup ( each 5 ml contain 640 mg of high DHA Fish oil) so we will give it in a dose 2.7 ml twice daily for children between 1 and 3 years and 3.5 ml twice daily for children between 4 and 5 years.
  Arms: Children with Pneumonia in intensive care unit receiving fish oil and the standard treatment

SUMMARY:
The aim of study is to investigate the effect of enteral feeding of Omega-3 on the outcome of children with Pneumonia in PICU

DETAILED DESCRIPTION:
Group A(cases) will be supplemented by omega-3 fatty acids for immediate post admission consecutive 7 days besides conventional treatment of pneumonia, in a dose of 350 mg twice daily for children less than 3 years and 450 mg twice daily for older children according to the standard treatment per the American Institute of Medicine of the National Academies guidelines for maximum dose for this age group. (Institute of Medicine of the National Academies,2016)

Side effects of omega-3 supplements are usually mild. They include unpleasant taste, bad breath, bad-smelling sweat, headache, and gastrointestinal symptoms such as heartburn, nausea, and diarrhea. (Office of Dietary Supplements ,2016)

Group B(controls) will be received enteral feeding without omega-3 fatty acid support.

ELIGIBILITY:
Inclusion Criteria

* All children patients with severe pneumonia admitted to PICU
* Both sexes
* Age: under 5 years
* Whose parents or caregivers approve for participation in the study

Exclusion Criteria

* Patients with chronic illnesses to exclude bias that could be emerged due to the chronic disease effect
* Whose parents or caregivers will not apply for participation in the study
* Patients who will be contraindicated for enteral feeding

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Hospital length stay | Through study completion, an average of 1 yea
  Hospital length stay will be measured between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hoda Atef Abdelsattar Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No